CLINICAL TRIAL: NCT06168929
Title: Bioequivalence Study of 2 Sizes of SHR4640 Tablets in Healthy Subjects (Randomized, Open, Single Dose, Two Sequences, Two Cycles, Self-Crossover Control)
Brief Title: Bioequivalence Study of 2 Sizes of SHR4640 Tablets Orally in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR4640-112
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — ruzinurad

STUDY DESIGN:
Intervention Model Description: Randomized, Open, Single Dose, Two Sequences, Two Cycles, Self-Crossover Control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR4640
- Treatment group B (Experimental)
  Interventions: Drug: SHR4640

INTERVENTIONS:
Drug: SHR4640 — SHR4640, 2.5mg*4 - 10mg*1
  Arms: Treatment group A
Drug: SHR4640 — SHR4640, 10mg*1 - 2.5mg*4
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the pharmacokinetic, and safety of two sizes of SHR4640 tablets in healthy adults, to explore the bioequivalence between two sizes of SHR4640 tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. 18 years to 45 years (inclusive).
3. Body weight should above 45 kg, and body mass index should be between 19 and 28 kg/m2 (inclusive).
4. The physical examination, vital signs, laboratory examination and electrocardiogram are not abnormal or abnormal but with no clinical significance.

Exclusion Criteria:

1. Pregnant or nursing women.
2. No birth control 1 weeks before screening or until one week after SHR4640 administration.
3. Average daily alcohol consume more than 14g for female or more than 28g for male within 1 month before screening, or baseline alcohol screening is positive.
4. Smokers (average daily smoking of 5 cigarettes or more in the 3 months before screening).
5. Subject with a history of substance abuse and drug abuse.
6. The investigators determined that other conditions were inappropriate for participation in this clinical trial.
7. sUA level ≥480 μmol/L.
8. eGFR < 90 mL/min/1.73 m2.
9. Positive result for human immunodeficiency virus (HIV), hepatitis C virus antibody, or syphilis antibody, or hepatitis B surface antigen.
10. 12-lead electrocardiogram (ECG) showed abnormal and clinically significant.
11. Cardiovascular, neuropsychiatric, respiratory, digestive tract, endocrine and other systemic diseases within 1 year before screening, which were judged to be serious by the investigators.
12. History of hypersensitivity to SHR4640 or its analogues.
13. History or suspected crystals or stones in the urinary system during the screening period of B-ultrasound.
14. History of been diagnosed with acute kidney injury in the past or screening period.
15. Had undergone major surgery within 3 months prior to screening, or have not recovered from surgery, or plan major surgery during the study.
16. Blood donation within 1 month before screening; Or patients with trauma or major surgical procedures who donated blood or lost blood > 400 mL in the 3 months prior to screening.
17. Has unsuitable venous for blood sampling.
18. Received the last dose of a study drug (or treatment with a medical device) within 3 months or 5 T1/2 (whichever is longer) of the screening or are currently participating in another study of a study drug (or medical device).
19. Have received or been exposed to other live vaccines or live attenuated vaccines within 3 months prior to Day 1, or who plan to receive live vaccines or live attenuated vaccines during the study.
20. Consumes grapefruit and/or poppy seed within 48 hours before SHR4640 administration.
21. Taken any prescription drugs, over-the-counter drugs, herbal medicines or food supplements within 2 weeks before screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
PK parameters of SHR4640: Cmax | 0 hour to 72 hour after administration
PK parameters of SHR4640: AUC0-t | 0 hour to 72 hour after administration
PK parameters of SHR4640: AUC0-inf | 0 hour to 72 hour after administration

SECONDARY OUTCOMES:
PK parameters of SHR4640: Tmax | 0 hour to 72 hour after administration
PK parameters of SHR4640: t1/2 | 0 hour to 72 hour after administration
PK parameters of SHR4640: CL/F | 0 hour to 72 hour after administration
PK parameters of SHR4640: Vz/F | 0 hour to 72 hour after administration
Adverse events | from ICF signing date to approximate day 13

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital Affilated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided